CLINICAL TRIAL: NCT06091735
Title: A Single-center, Single-blind, Randomized Controlled Clinical Study of Bowel Preparation Before Colonoscopy
Brief Title: Clinical Study of Bowel Preparation Before Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Shupei Li, student, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DZQH-KYLL-23-11
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Magnesium sulfate sodium potassium solution group (Experimental): Magnesium sulfate sodium potassium solution group: 3L magnesium sulfate sodium potassium oral concentrated solution. At 18:00 1d before the inspection, dissolve a package of contents into 200ml with water, and drink 250ml of water every half hour after that, drinking a total of 6 cups (that is, 1.5L); On the day of the examination (6 hours before the colonoscopy) repeat the same medication as the previous evening.
  Interventions: Drug: OSS
- Magnesium sulfate sodium potassium solution group + linaclotide group (Experimental): Magnesium sulfate sodium potassium solution + linaclotide group: 3L sodium magnesium sulfate potassium oral concentrated solution + linaclotide 290μg. One tablet of linalotide was taken orally at 18:00 one day before the examination, and then two packets of contents were dissolved into 300ml with water 6 hours before the colonoscopy. After that, 500ml of water was drunk every half hour, for a total of 6 cups.
  Interventions: Drug: OSS+Linzess
- PEG (Compound polyethylene glycol electrolyte powder) group (Placebo Comparator): PEG (Compound polyethylene glycol electrolyte powder) group: 3LPEG. At 18:00 1d before the inspection, dissolve a package of contents into 200ml with water, and drink 250ml of water every half hour after that, drinking a total of 6 cups; On the day of the examination (6 hours before the colonoscopy) repeat the same medication as the previous evening.
  Interventions: Drug: PEG-Interferon Alfa

INTERVENTIONS:
Drug: OSS — experimental
  Other Names: Sodium potassium magnesium sulfate oral concentrated solution
  Arms: Magnesium sulfate sodium potassium solution group
Drug: OSS+Linzess — experimental
  Other Names: sodium potassium magnesium sulfate oral concentrated solution + linaclotide
  Arms: Magnesium sulfate sodium potassium solution group + linaclotide group
Drug: PEG-Interferon Alfa — Placebo Comparator
  Other Names: PEG
  Arms: PEG (Compound polyethylene glycol electrolyte powder) group

SUMMARY:
This study was a single-center, randomized controlled clinical study. Subjects meeting the inclusion criteria will be randomly assigned to magnesium sodium potassium sulfate oral concentrated solution group, magnesium sodium potassium sulfate oral concentrated solution + linaclotide group, PEG group in equal proportion.

DETAILED DESCRIPTION:
Research purpose

In this study, by evaluating patients' intestinal cleanliness rate (BBPS score) and quantitative analysis of intestinal bubble under colonoscopy, three intestinal preparation schemes were respectively investigated: The effectiveness, tolerability, adverse reactions and prognosis of concentrated oral solution of sodium and potassium magnesium sulfate (experimental group 1), concentrated oral solution of sodium and potassium magnesium sulfate + linalotide (experimental group 2), PEG(compound polyethylene glycol electrolyte powder) (control group) were analyzed and compared, in order to improve the intestinal preparation cleanliness rate of colonoscopy subjects.

3. Study the overall design

1. Research program design A single-center, single-blind, randomized controlled parallel design was adopted.
2. Entry criteria Patients aged ≥18 years and ≤80 years who need intestinal preparation before colonoscopy.
3. Study sample size In this study, PASS 15 software was used to estimate the sample size. According to previous research data, the intestinal cleanliness rates of the three groups of sodium and potassium magnesium sulfate oral concentrated solution group (test group 1), sodium and potassium magnesium sulfate oral concentrated solution + linalotide group (test group 2) and PEG group (control group) were set to be 86%, 90% and 69.36%, respectively, and the differences between the two groups and the control group were mainly compared. Considering that the total Class I error rate of multiple tests is controlled within 0.05, the bilateral test level of both tests is set as α=0.025, and the degree of assurance is 80%, and the minimum sample size of each group is calculated as 118 cases according to the equal ratio of 1:1:1. Considering a possible 20% shedding rate, it is planned to include 148 patients in each group, for a total of 444 patients.
4. Criteria for judging clinical efficacy 4.1 Main therapeutic indexes Evaluation criteria for the main efficacy indicators: The proportion of subjects with a total Boston score ≥6 and a colon score ≥2 for each segment was recorded as effective.

the Boston bowel preparation scale (BBPS) can be used to evaluate the volume, morphology and mucosal clarity of stool and fluid in the bowel. The scoring criteria are as follows: 0 points: there is stool in the colon that cannot be cleared, and the mucosa can not be seen clearly, which is mostly seen in the stage without intestinal preparation;

1. Part of the intestinal mucosa was clearly displayed, while the other part of the mucosa was not clearly displayed due to feces and opaque liquid residues; 2 points: There is a small amount of stool and opaque liquid remaining in the colon; 3 points: All mucous membranes are clearly displayed, and no stool or opaque fluid remains in the colon.

Rating description:

1. The colon score of each segment was 0~3, and the total score was 0~9:
2. The colon score of each segment was ≥2, indicating adequate intestinal preparation:
3. The total score of 6 and the score of any segment of colon < 2 were classified as inadequate intestinal preparation.
4. The total score ≥6 and the colon score ≥2 points in each segment indicated that the intestinal preparation was adequate, otherwise it was inadequate.

   4.2 Secondary efficacy indicators Evaluation criteria of secondary curative effect indicators: those who scored 1 or 2 points (i.e., > 0 points) under colonoscopy were recorded as satisfied.

   Colonoscopic evaluation of intestinal bubbles, the scoring criteria are as follows:

0 points: there are many bubbles in the intestinal cavity, requiring a lot of water to rinse repeatedly after observation;

1 point: there are few bubbles in the intestinal cavity, which need to be observed after a small amount of washing; 2 points: There are almost no bubbles in the intestinal cavity, and it can be observed well without rinsing.

4. Case selection

1. Study subjects: patients aged ≥18 years and ≤80 years who need intestinal preparation before colonoscopy.
2. Inclusion criteria:

1) Signed written informed consent; 2) Age 18-80 years old, gender is not limited; 3) The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale; 4) Non-lactating pregnant women and no pregnancy plan during the test; 5) Do not participate in any clinical trials for 3 months before and during the trial; 6) Participate voluntarily and sign informed consent. 3. Exclusion criteria

1. NYHA cardiac function grade III or IV;
2. Unstable angina pectoris in the convalescence period of acute myocardial infarction or in the near future;
3. have serious liver and kidney function diseases;
4. Suspected gastrointestinal obstruction or gastrointestinal perforation;
5. Pregnant or lactating women;
6. Mental illness or physical dysfunction can not cooperate with the examination;
7. People who are allergic to intestinal preparation drugs.
8. Patients who did not undergo colonoscopy after bowel clearing due to their own reasons;
9. Patients who can not tolerate general colonoscopy and terminate the examination;
10. Patients who requested withdrawal from the study. 5. Clinical trial procedures

<!-- -->

1. Overview: The subjects signed informed consent and were randomly assigned to complete intestinal preparation according to the requirements of the corresponding drugs, and underwent colonoscopy and routine postoperative treatment. The subjects were asked to receive regular telephone follow-up or outpatient follow-up, receive recent information, imaging examination, laboratory examination and other methods to evaluate the effects of the drugs, collect complete medical records and complete statistics.
2. Treatment grouping and random allocation:

   In this study, biostatistics professionals used the block randomization method with variable block length to generate a random assignment sequence, and the enrolled subjects were randomly assigned to three groups in equal proportion (1:1:1). The three treatment groups were: (1) sodium and potassium magnesium sulfate solution group: 3L oral concentrated solution of sodium and potassium magnesium sulfate. At 18:00 1d before the inspection, dissolve a package of contents into 200ml with water, and drink 250ml of water every half hour after that, drinking a total of 6 cups (that is, 1.5L); On the day of the examination (6 hours before the colonoscopy) repeat the same medication as the previous evening. (2) Magnesium sulfate sodium potassium solution + linaclotide group: 3L sodium magnesium sulfate potassium oral concentrated solution + linaclotide 290μg. One tablet of linalotide was taken orally at 18:00 one day before the examination, and then two packets of contents were dissolved into 300ml with water 6 hours before the colonoscopy. After that, 500ml of water was drunk every half hour, for a total of 6 cups. (3) PEG (Compound polyethylene glycol electrolyte powder) group: 3LPEG. At 18:00 1d before the inspection, dissolve a package of contents into 200ml with water, and drink 250ml of water every half hour after that, drinking a total of 6 cups; On the day of the examination (6 hours before the colonoscopy) repeat the same medication as the previous evening.

   In practice, the mobile phone-based "Ratjin" wechat mini program was used to achieve random allocation of the three treatment groups (the specific randomization scheme will be developed separately). When the subjects sign the informed consent, and the subjects meeting the test enrollment conditions need to be randomized after screening, the authorized researcher will input the relevant information of the patients in the mobile phone client, and after the approval and confirmation of the designated random administrator, the assigned group will be immediately fed back to the mobile phone, and the researcher will implement the corresponding treatment for the patients according to the randomly assigned group. This method can generate random assignment sequence in advance, realize random assignment concealment completely, and prevent selection bias effectively.
3. Preparation before treatment: 2 days before colonoscopy, the three groups were forbidden to eat high-fiber vegetables, dragon fruit and other seeded fruits, and should mainly eat low-fiber and low-residue foods, and eat dinner before 6 PM, and then fast; Check for semi-liquid or liquid food the night before, and check for fasting and no drinking on the day.
4. Post-treatment: In order to replace fluid loss during the examination, the patient subsequently drinks an adequate amount of fluid to maintain adequate hydration. Seek medical attention if severe or persistent diarrhea occurs.
5. Participants in the test and division of labor 1) 3 experienced endoscopists and several experienced endoscopic nurses cooperated with the doctor to complete the use of endoscopic instruments.

2) 2 researchers observed and recorded, and carried out related work: A. After colonoscopy, the researchers recorded and statistically analyzed the intestinal cleanliness of the subjects, the content of bubbles in the intestinal cavity, the location, size and number of detected polyps, and adenomatous polyps.

B. Record, observe and record the occurrence of adverse reactions (such as the occurrence of nausea, vomiting, headache, dizziness, abdominal pain, abdominal distension, etc.); C. Assist with various incidents. 6. Follow-up procedure Observation node and follow-up procedure: After colonoscopy, the patients were asked about their satisfaction with the taste of laxatives, whether they were satisfied with this group of bowel cleansing methods, adverse reactions (nausea, vomiting), etc.

7. Observation indicators

1. General information: age, sex, ethnicity, occupation, height, weight, medical history, medication history, contact address and telephone number
2. Main outcome measures: Patients' intestinal cleanliness rate (BBPS score).
3. Secondary observation indicators: The evaluation of intestinal bubble under colonoscopy, the detection rate of adenoma, the detection rate of polyps, the admission time, exit time and total colonoscopy time of the patients, the actual drug tolerance and satisfaction of the subjects, the amount of exercise, the speed and time of exercise, the amount of water they drank, whether they had colonoscopy for the first time, whether they were usually constipation, and the reasons for colonoscopy of the patients were observed. Patients' satisfaction with education methods and the occurrence of adverse reactions. Blood routine, urine routine, stool routine, coagulation function, blood biochemistry, etc.
4. Other biological indicators: body temperature, heart rate, respiration, blood pressure, etc.
5. Safety indicators: blood routine, urine routine, stool routine, coagulation function, biochemistry, adverse reactions.

8. Exit indication

Subjects may withdraw from the study at any time if:

1. The subject voluntarily withdraws the informed consent; 2. Subjects with adverse reactions or serious adverse reactions; 3. Subjects have poor compliance and do not follow medical advice; 4. Natural shedding. 9. Statistical methods

1. Analyze the data set Three data analysis sets were used for statistical analysis: full analysis set (FAS), conformance scheme set (PPS) and security analysis set (SS). FAS will serve as the data set for baseline and primary efficacy measures analysis, PPS for all efficacy measures analysis, and SS for safety analysis. FAS included all participants who met the inclusion criteria to enter the study, received the necessary treatment, and had at least one follow-up evaluation of efficacy; Patients who seriously violated the exclusion criteria and did not have any follow-up data after enrollment were excluded. PPS included all subjects that met the admission criteria, completed all follow-up according to protocol requirements, had no major protocol violations, and had good compliance. SS included all participants who entered the study, received the necessary treatment, and were followed up for safety evaluation.

   When FAS is used for analysis, the missing data of the main efficacy indicators will be analyzed after data filling in a relatively conservative method according to the specific situation, and sensitivity analysis will be performed if necessary. Other indicators will not be filled with missing data.
2. Statistical analysis methods In this study, SAS 9.4 software was used for statistical analysis.

1) Descriptive statistics Different statistical indicators were adopted according to the type of variables. Continuous variables were described by mean, standard deviation, median, and upper and lower quartiles. The categorical variables were described by frequency and percentage.

2) Difference test The comparison among the three groups of continuous variables with the same variance and normal distribution was conducted by One-way ANOVA, and Welch calibration test was used when the variance was inconsistent. The Kruskall-Wallis H test was used to compare the three groups of continuous variables that do not obey normal distribution. Comparisons between groups of categorical variables were performed using Pearson Chi-square test or Fisher exact probability test. P≤0.05 was defined as a statistically significant difference. If further pairwise multiple comparisons are required, Bonferroni correction is used.

3) Main therapeutic indexes The main outcome indicators of patients' intestinal cleaning rate (BBPS score) and colonoscopic enteric bubble evaluation were compared between two groups (magnesium sodium potassium solution group vs. PEG group, magnesium sodium potassium solution + linalotide group vs. PEG group) using Pearson Chi-square test, P≤0.025 was defined as statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Age 18-80 years old, gender is not limited;
* The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale;
* Non-lactating pregnant women and no pregnancy plan during the test;
* Do not participate in any clinical trials for 3 months before and during the trial;
* Participate voluntarily and sign informed consent.

Exclusion Criteria:

* NYHA cardiac function grade III or IV;
* Unstable angina pectoris in the convalescence period of acute myocardial infarction or in the near future;
* have serious liver and kidney function diseases;
* Suspected gastrointestinal obstruction or gastrointestinal perforation;
* Pregnant or lactating women;
* Mental illness or physical dysfunction can not cooperate with the examination;
* People who are allergic to intestinal preparation drugs.
* Patients who did not undergo colonoscopy after bowel clearing due to their own reasons;
* Patients who can not tolerate general colonoscopy and terminate the examination;
* Patients who requested withdrawal from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
BBPS | 1day
  The proportion of subjects with an overall Boston score ≥6 and a colon score ≥2 for each segment was considered valid.

CONTACTS AND LOCATIONS:
Locations (1):
- A single-center, single-blind, randomized controlled clinical study of bowel preparation before colonoscopy, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No